CLINICAL TRIAL: NCT05390164
Title: Sensory Symptoms as an Early Manifestation of Active Vitiligo: a Case-control Clinical and Molecular Study
Brief Title: Sensory Symptoms in Active Vitiligo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Other Study IDs: Pruritis in vitiligo
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Totest Sensory Symptoms in Active Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active vitiligo
  Interventions: Diagnostic Test: skin biopsy
- Stable vitiligo
  Interventions: Diagnostic Test: skin biopsy

INTERVENTIONS:
Diagnostic Test: skin biopsy — skin biopsy to be analyzed by ELISA

SUMMARY:
This work aims to assess sensory symptoms in early active vitiligo patients (segmental, non-segmental, or mixed) and to measure 3 neuropeptides expression in their lesional skin [neuropeptide Y(NPY), calcitonin gene-related peptide (CGRP), and nerve growth factors (NGF)] to correlate neuropeptide levels, sensory symptoms, and functions, with criteria of disease activity and perceived stress scale.

DETAILED DESCRIPTION:
Study Design: Case-control study Population: 45 patients with active vitiligo and 45 patients with stable vitiligo

Inclusion criteria:

Age: 18 years old and older Sex: both sexes

Exclusion criteria:

Other hypopigmented diseases such as pityriasis alba, tinea versicolor, lichen sclerosis, post-inflammatory hyperpigmentation, and leprosy as excluded by lack of accentuation by wood's light examination. - Cases who received treatment (systemic or topical) in the last 3 months before sampling. - Neurological or other diseases that cause itching. - Medical history of DM, HTN, or other systemic diseases, history of associated autoimmune diseases.

Assessment will be carried as follows: • History of itching or other abnormal neurological sensations as paresthesia and numbness. Aggravating factors (e.g. dryness, hot environment, sun exposure, ..etc), alleviating factors of itching Type of vitiligo (segmental, unilateral, vulgaris). • Assessment of activity by assessing: koebner's phenomenon, confetti depigmentation, trihypochrome areas, poorly defined borders, inflammatory signs (e.g eye inflammation and hearing loss), and leukotrichia. • Assessment of sensory symptoms and signs (fine touch, crude touch, pain, and sweating by starch iodine test) in active vitiliginous patches. • Clinical assessment: the vitiligo area score index (VASI), vitiligo extent scores (VES), vitiligo disease activity score (VIDA) (Feily, 2014) will be assessed in every participant and demographic data

ELIGIBILITY:
Inclusion Criteria:

* Active and stable vitiligo

Exclusion Criteria:

* Diabetic or other associated disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Active vitiligo patients
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Neuropeptide | 3 months
  laboratory test

REFERENCES:
- [Derived] El Sayed H, El Wakeel H, Nour Z, Mohyeeldeen R, Hafez V. Sensory Symptoms as an Early Manifestation of Active Vitiligo: A Case-Control Clinical and Molecular Study. Pigment Cell Melanoma Res. 2025 Jan;38(1):e13223. doi: 10.1111/pcmr.13223. PMID 39869070